CLINICAL TRIAL: NCT02618070
Title: Cognitive Modulation of Dyspeptic Symptom During Food Ingestion in Functional Dyspepsia Patients Cognitive Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Inseon Lee, MS, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 633/2015BO2
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Brain Imaging; Functional Dyspepsia; Food
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Functional dyspepsia patient (Experimental): Yogurt ingestion
  Interventions: Other: Yogurt
- Healthy (Experimental): Yogurt ingestion
  Interventions: Other: Yogurt

INTERVENTIONS:
Other: Yogurt

SUMMARY:
In this functional magnetic resonance imaging study, effects of different information of fat content of high or low fat will be examined in FD patients and healthy volunteers (n=30, respectively). These data will provide a better understanding of symptom generation following food ingestion in general as well as in patients with respective functional gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, volunteering adults BMI: 18-25 kg/m² right-handed Age: 18-65 years Capacity to give informed consent

For FD patients, Diagnosis of functional dyspepsia over the last 12 months certified by a medical record Inconspicuous gastroscopy during the last 6 months certified by a medical record

Exclusion Criteria:

* Subjects which have a non-removable metal object in or at their body, such as, for example:
* Heart pace-maker,
* Artificial heart valve,
* Metal prosthesis,
* Metallic implants (screws, plates from operations, etc.),
* Interuterine Spiral,
* Metalsplinters / grenade fragments
* Non-removable dental braces,
* Acupuncture needles,
* Insulin pump,
* Intraport, etc., Pregnant women or pregnancy cannot be excluded Nursing women Subjects with limited temperature perception and/or increased sensitivity to warming of the body A circulatory disease cannot be excluded Subjects with hearing-disease or an increased sensitivity to loud noises Subjects with fear of closed-in places (claustrophobia) Subjects which were operated less than three month ago Acute illness or infection Neurological disorder or injury (e.g. epilepsy) Moderate or severe head injury Severe psychotic illness (e.g. schizophrenia, depression) Intake of antidepressants / antipsychotics Vegetarians/Vegans Food allergies Self-reported eating disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
functional brain activity | 1-2 years
  Resting BOLD (Blood oxygenation level-dependent) signal before and after yogurt ingestion will compared between groups.
  There is a small risk of discomfort from claustrophobia, periods of immobility, and exposure to the noise of the magnet. The investigators will offer the participants ear plugs. In rare cases the participants experience dizziness, nausea, or tinnitus which normally disappear after the measurement. During the measurements there is the possibility of warming which could lead to skin irritation in people with tattoos. Therefore, the participants with tattoos will not be included. The participants are instructed to tell the investigators immediately if any uncomforted appears. The study will be performed by experienced experimenters who know all about the risks. During the measurements, the participants are monitored. As a commercial yogurt (200 ml) will be used, the investigators do not expect any side effects. Food allergy will be checked before.
subjective rating | 1-2 years
  The investigators will measure how much the participants have fullness, satiation, nausea and vomiting, pain, and their mood before and after the yogurt ingestion using visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Enck, Prof., Principal Investigator — Psychosomatic Medicine and Psychotherapy Department, University of Tübingen, Tübingen, Germany
Locations (1):
- Psychosomatic Medicine and Psychotherapy Department, University of Tübingen, Tübingen, Germany, Tübingen, Germany

REFERENCES:
- [Derived] Lee IS, Kullmann S, Scheffler K, Preissl H, Enck P. Fat label compared with fat content: gastrointestinal symptoms and brain activity in functional dyspepsia patients and healthy controls. Am J Clin Nutr. 2018 Jul 1;108(1):127-135. doi: 10.1093/ajcn/nqy077. PMID 29924294